CLINICAL TRIAL: NCT04975646
Title: Goal Attainment Scaling in Upper Limb Spasticity Treatment With Botulinum Toxin and the Influence of Regular Exercise for Spastic Upper Limb on Quality of Life in Patients After Stroke
Brief Title: Goal Attainment Scaling in Upper Limb Spasticity Treatment
Acronym: GASBTX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Rehabilitation Institute, Republic of Slovenia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202102
Record Dates: First submitted 2021-02-15; First posted 2021-07-23 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Ischemic Stroke; Hemorrhagic Stroke
Keywords: rehabilitation; spasticity; botulinum toxin A; goal setting; spasticity-related quality of life
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke; Muscle Spasticity

STUDY DESIGN:
Intervention Model Description: First part: observational study. Second part: parallel groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Prescribed exercise program
  Interventions: Behavioral: Prescribed exercise program
- Control group (No Intervention): Exercising at patient's own discretion

INTERVENTIONS:
Behavioral: Prescribed exercise program — Active or passive exercises for the spastic upper limb, including functional electrical stimulation (FES), performed regularly for two weeks.
  Arms: Test group

SUMMARY:
Patients after stroke with upper limb spasticity treated with botulinum toxin-A (BTX-A) will be included in this two-part study. In the first part, goal attainment scaling and comprehensive assessment of motor functioning will be performed before BTX-A application and after two weeks. In the second part, the patients will be randomised into a test group performing prescribed regular exercise for two weeks and a control group exercising at their own discretion during the same period, whereby the patients' health-related quality of life will be assessed at the beginning and end of the two-week period.

DETAILED DESCRIPTION:
Goal setting will be performed by the patient together with the physician according to the SMART principle (specific, measureable, achievable, realistic, time bound). The goals will be classified according to the International Classification of Functioning, Disability and Health. Goal attainment will be assessed using the Goal Attainment Scale - Light. Comprehensive assessment of motor functioning will address range of motion, spasticity, pain, degree of motor disability and degree of dependence in daily activities. The prescribed exercises for the test group will be passive or active, depending on spasticity of the impaired upper limb. Both groups will keep an Exercise Diary during the second part of the study.

ELIGIBILITY:
Inclusion Criteria:

* patient's or caregiver's approval
* ischemic or hemorrhagic stroke diagnosed using head CT/MRI
* at least one upper limb muscle spasticity (MAS ≥ 3)
* candidate for BTX-A treatment or already given BTX-A in the past
* patient's or caregiver's capability for goal attainment protocol cooperation (Mini Mental Examination ≥ 24 points)

Exclusion Criteria:

* aphasic patients without caregiver's presence
* other neurological or musculoskeletal diseases that could affect the treatment outcome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-01-03 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
GAS-Light | At baseline, after 2 weeks (i.e., at the end of the 1st part of the study)
  Change in Goal Attainment Scale - Light
SQoL-6D | Start of the 2nd part of the study (i.e., after 2 weeks), end of the 2nd part of the study (i.e., after 4 weeks)
  Change in Spasticity Related Quality of Life Tool score

SECONDARY OUTCOMES:
ROM | Start of the 2nd part of the study (i.e., after 2 weeks), end of the 2nd part of the study (i.e., after 4 weeks)
  Change in Range of motion (degrees)
MAS | Start of the 2nd part of the study (i.e., after 2 weeks), end of the 2nd part of the study (i.e., after 4 weeks)
  Change in Modified Ashworth Scale score
PSFS | Start of the 2nd part of the study (i.e., after 2 weeks), end of the 2nd part of the study (i.e., after 4 weeks)
  Difference in Penn Spasm Frequency Scale
VAS | Start of the 2nd part of the study (i.e., after 2 weeks), end of the 2nd part of the study (i.e., after 4 weeks)
  Change in pain rating on the Visual Analog Scale
BSR | Start of the 2nd part of the study (i.e., after 2 weeks), end of the 2nd part of the study (i.e., after 4 weeks)
  Change in Brunnstrom Stage of Recovery score
MRS | Start of the 2nd part of the study (i.e., after 2 weeks), end of the 2nd part of the study (i.e., after 4 weeks)
  Change in Modified Rankin Scale score

CONTACTS AND LOCATIONS:
Overall Officials: Nataša Bizovičar, MD, PhD, Principal Investigator — University Rehabilitation Institute, Republic of Slovenia
Locations (1):
- University Rehabilitation Institute, Republic of Slovenia, Ljubljana, Slovenia